CLINICAL TRIAL: NCT07333157
Title: Effects of Wearable Passive Back Support Suit on Back Pain in Caregivers
Acronym: back pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Won Hyuk Chang, professor, Samsung Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-01-010
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Back Pain; Exoskeleton Device
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- wearable passive back support suit (Experimental)
  Interventions: Device: wearable passive back support suit
- traditional lumbosacral orthosis (Active Comparator)
  Interventions: Device: traditional lumbosacral orthosis

INTERVENTIONS:
Device: wearable passive back support suit — 2-week intervention periods using a wearable passive back support (Angel GEAR soft B10, Angel Robotics, Co., Ltd)
  Arms: wearable passive back support suit
Device: traditional lumbosacral orthosis — 2-week intervention periods using a traditional lumbosacral orthosis.
  Arms: traditional lumbosacral orthosis

SUMMARY:
The physical demands of patient transport, including lifting and transferring patients, are significant contributors to the high risk of musculoskeletal disorders. Previous studies have demonstrated that these workers frequently experience musculoskeletal pain. Although current prevention strategies primarily consist of passive education on posture, there is a clear need for more active, assistive methods. The emergence of wearable passive back support suits as a potential solution is noteworthy; however, robust clinical research on the effectiveness of these devices in real-world care giving environments is currently lacking.

The objective of this study is to investigate the effects of a wearable passive back support suit on reducing and preventing the incidence of back pain in patient transporters.

ELIGIBILITY:
Inclusion Criteria:

1. Male adults aged 19 years or older
2. Patient transport staff at Samsung Medical Center
3. Able to wear a wearable passive back support suit

   * Height: 156cm-188cm
   * Chest circumference: 80cm-120cm
   * Thigh circumference: 36cm-62cm

Exclusion Criteria:

1. Severe musculoskeletal disorders of the spine
2. Severe musculoskeletal disorders of the lower extremities
3. Contractures limiting the range of motion of the spine and lower extremities
4. Fractures, open wounds, or unhealed ulcers on the spine or lower extremities
5. Difficulty using a lumbar support device due to severe medical conditions, such as cardiovascular or pulmonary diseases
6. History of osteoporotic fractures
7. Neurological disorders affecting gait (e.g., stroke, Parkinson's disease, multiple sclerosis, etc.)
8. Any other cases where the investigator determines that participation in this study is inappropriate

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-03-21 (Actual); Primary Completion 2025-07-24 (Actual); Study Completion 2025-07-24 (Actual)

PRIMARY OUTCOMES:
Change in the Korean Oswestry Low Back Pain Disability Questionnaire(K-ODI) score | baseline, Week 2(after period 1), week 4(after washout) and week 6 (after period 2)

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea